CLINICAL TRIAL: NCT04538677
Title: Video Consultation During Follow up Care: Effect on Quality of Care and Patient- and Provider Attitude in Patients With Colorectal Cancer
Brief Title: Video Consultation During Follow up Surgical Care
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof. dr. W.A. Bemelman, Prof. dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: W17_149
Record Dates: First submitted 2020-08-31; First posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: Colorectal Cancer
Keywords: Video Consultation; Virtual visits
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- F2F-Group: Patients who preferred a traditional F2F-appointment were seen at the outpatient clinic.
- VC-group: Patients who preferred a video consult were seen over a video connection.
  Interventions: Device: Video consultation

INTERVENTIONS:
Device: Video consultation — A two-way audio and visual connection between patients and surgeons
  Groups: VC-group

SUMMARY:
The aim of this study was to compare the willingness to use and attitude towards VC amongst both patients with colorectal cancer and healthcare providers during follow up care. Second, to determine the satisfaction with the quality of the healthcare provider and the usability of the used VC technology. 50 patients will be asked to choose between video consultation or face-to-face contact at the outpatient surgical clinic.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Fluent in speaking and writing in Dutch
* Follow up appointments in which overall progress, new complaints, results with good news and treatment was discussed were considered feasible.

Exclusion Criteria:

* Introductory appointments
* Bad news consultations
* Physical examination needed
* No access to Internet
* No access to a smartphone, tablet or computer with a camera
* Not willing to activate their electronic patient portal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colorectal cancer scheduled for appointment at the surgical oncology outpatient a tertiary referral center.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-08-23 (Actual); Study Completion 2017-08-23 (Actual)

PRIMARY OUTCOMES:
Attitude and satisfaction with video consultation | Immediately after the consult
  PAT-VC questionnaire

SECONDARY OUTCOMES:
Usability of the video consultation technology | Immediately after the test consult
  SUS questionnaire
Quality of provided care by surgeon: MSF questionnaire | Immediately after the consult
  MSF questionnaire
Satisfaction of surgeons: Questionnaire | Immediately after the consult
  Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, location AMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR